CLINICAL TRIAL: NCT05042414
Title: Acute Effects of Endurance Exercise on Breastmilk Composition: Pilot Study
Brief Title: Acute Effects of Endurance Exercise on Breastmilk Composition
Acronym: ExMilk
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Basic Science
Other Study IDs: 263493
Record Dates: First submitted 2021-08-13; First posted 2021-09-13 (Actual); Last update posted 2022-10-10 (Actual); Status verified 2022-10

CONDITIONS: Breastmilk
Keywords: Exercise
MeSH Terms: conditions — Motor Activity | interventions — High-Intensity Interval Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Breastmilk (Experimental): Randomized intervention order.
  Interventions: Behavioral: High intensity interval training; Behavioral: Moderate intensity training; Behavioral: Resting

INTERVENTIONS:
Behavioral: High intensity interval training — Four times four minutes treadmill interval training
Behavioral: Moderate intensity training — Moderate intensity treadmill training
Behavioral: Resting — No training

SUMMARY:
The investigators will determine the acute effect of exercise on breastmilk composition. Participants will come in to the lab on three different days, out of which they will exercise on two of these days and rest in the lab on the third day. The conditions will be randomly allocated to each participant. Breastmilk samples will be obtained in the morning of each test day, as well as immediately after, one hour after and four hours after the exercise/rest condition. Dietary intake will be standardized on the test days. At the time of study commencement, the trial (including planned analyses) is not fully funded. Additional milk will be stored for future analyses (not yet specified) when funding is secured.

ELIGIBILITY:
Inclusion Criteria:

* 6 to 12 weeks postpartum
* Exclusive breastfeeding
* Term birth

Exclusion Criteria:

* Known cardiovascular disease
* Type 1 or 2 diabetes mellitus
* Limited ability to exercise

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2021-08-24 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2022-06-01 (Actual)

PRIMARY OUTCOMES:
Breastmilk metabolite composition | Change from before exercise to after exercise (+0 hour, +1 hour, and + 4 hours)
  Metabolomics profiling

SECONDARY OUTCOMES:
Adiponectin | Change from before exercise to after exercise (+0 hour, +1 hour, and + 4 hours)
  Concentration in breastmilk
Leptin | Change from before exercise to after exercise (+0 hour, +1 hour, and + 4 hours)
  Concentration in breastmilk
Insulin | Change from before exercise to after exercise (+0 hour, +1 hour, and + 4 hours)
  Concentration in breastmilk
Insulin Growth Factor-1 | Change from before exercise to after exercise (+0 hour, +1 hour, and + 4 hours)
  Concentration in breastmilk
Cytokine profiling (Multiplex 27) | Change from before exercise to after exercise (+0 hour, +1 hour, and + 4 hours)
  Concentration in breastmilk

OTHER OUTCOMES:
Cardiorespiratory fitness | At baseline
  Peak oxygen uptake
Body mass in kg | At baseline
  Impedance scale
Height in metres | At baseline
  stadiometer
Fat mass in kg | At baseline
  Impedance scale
Muscle mass in kg | At baseline
  Impedance scale

CONTACTS AND LOCATIONS:
Overall Officials: Øystein Risa, Phd, Study Director — Norwegian University of Science and Technology
Locations (1):
- Department of Circulation and Medical Imaging, NTNU, Trondheim, Norway

REFERENCES:
- [Derived] Lemoine MCC, Klau LJ, Holmen M, Ashby ER, Aachmann FL, Andreassen T, Giskeodegard GF, Moholdt T. Unaltered 3'-sialyllactose and 6'-sialyllactose concentrations in human milk acutely after endurance exercise: a randomized crossover trial. Front Nutr. 2025 Oct 27;12:1638430. doi: 10.3389/fnut.2025.1638430. eCollection 2025. PMID 41220705
- [Derived] Holm RL, Holmen M, Sujan MAJ, Giskeodegard GF, Moholdt T. Acute effect of endurance exercise on human milk insulin concentrations: a randomised cross-over study. Front Nutr. 2025 Jan 27;11:1507156. doi: 10.3389/fnut.2024.1507156. eCollection 2024. PMID 39981021